CLINICAL TRIAL: NCT01277796
Title: Pilot Study of Thermotherapy Treatment for Cutaneous Leishmaniasis in Peru With the HECT-CL Device
Brief Title: Pilot Study Using a Heat Pack to Treat Cutaneous Leishmaniasis
Acronym: HECT
Status: Available | Type: Expanded Access
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Tulane University School of Medicine (Other)
Responsible Party: Richard Witzig, MD, MPH, Associate Professor of Medicine., Infectious Diseases Section, Tulane School of Medicine.
Other Study IDs: 032-08
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous

INTERVENTIONS:
Device: Heat pack conduction-heat therapy — Hand warmer heat pack with reliable (and monitored) temperature (50-52 degrees Celsius) will be applied to lesion borders for 3 minutes (fractionated to 90 second intervals or less) every day, for 7 consecutive days.

SUMMARY:
Current standard therapies with chemotherapy (CT) for Cutaneous Leishmaniasis (CL) are expensive, toxic/allergenic, frequently ineffective, burdensome, and often unavailable. Thermotherapy is a clinically validated first line alternative for the treatment of Cutaneous Leishmaniasis in South America. However, current heat-delivery modalities are either too costly or lack governmental approval required to be made widely available to endemic areas. The investigators have adapted a reliable, safe, and low-cost heat pack for Cutaneous Leishmaniasis that the investigators have named the HECT-CL device. In this pilot study the investigators will enroll 25 patients who have either failed or are not candidates for pentivalent antimonies. The hypothesis states that the HECT-CL device demonstrates efficacy non-statistically inferior to estimates for current South American Pentavalent Antimonial cure rates (76%) while demonstrating basic safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* with CL diagnosed by skin smear (WHO method), biopsy, culture, PCR
* aged 8-80 years old
* with no more than 3 lesions
* ulcerative and non-ulcerative ulcers less than 4 cm diameter.
* allergy, prohibitive side effects to standard chemotherapy, or other contraindication to antimonial treatment (e.g. cardiac arrhythmia)
* capable of signing an informed consent or having capable guardians (in the case of minors).
* Children ≥ 8 years of age must give written or verbal informed assent along with written consent of their guardians.

Exclusion Criteria:

* lesions less than 2cm from the nose, mouth, ears, or eyes.
* clinically diagnosed with mucosal involvement.
* evidence of lymph node involvement on exam.
* unable or unwilling to commit to the treatment and follow-up plan.
* prior CL treatment within last 1 month.
* pregnant or lactating
* uncontrolled severe systemic illness or immunocompromised state.

Ages: 8 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Llanos-Cuentas, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Witzig Richard, MD, MPH, Principal Investigator — Tulane Medical School